CLINICAL TRIAL: NCT02154217
Title: Comparison of the Effects of Bimatoprost and a Fixed Combination of Latanoprost and Timolol on 24-hour Blood and Ocular Perfusion Pressures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Paolo Fogagnolo, MD, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LR-BLT
Record Dates: First submitted 2014-05-21; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Bimatoprost; Latanoprost; Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bimatoprost (Experimental): once daily
  Interventions: Drug: Bimatoprost
- Latanoprost/Timolol (Experimental): once daily
  Interventions: Drug: Latanoprost/Timolol

INTERVENTIONS:
Drug: Bimatoprost
  Arms: Bimatoprost
Drug: Latanoprost/Timolol
  Arms: Latanoprost/Timolol

SUMMARY:
This is a data revision with a focus on 24 hour perfusion pressures of data from a previous randomized, double masked, multicenter clinical trial.

The aim was to compare the effect of bimatoprost and the fixed combination of latanoprost and timolol (LTFC) on 24-hour mean intraocular pressure (IOP) after patients are switched from a nonfixed combination of latanoprost and timolol.

The main findings of the original trial had been published on Ophthalmology [2007;114: 2244-2251].

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed as having POAG (primary open-angle glaucoma) or ocular hypertension and 18 years or older who fulfilled the eligibility requirements detailed below and signed an informed consent at the screening visit were included.

Two different groups of patients were potentially eligible:

1. Those patients who were controlled (IOP< 21 mmHg) on the nonfixed combination of latanoprost and timolol (twice daily or once daily morning administration) for at least 3 months prior to the baseline visit.
2. Patients on monotherapy either with latanoprost or timolol who were eligible for dual therapy being not satisfactorily controlled (IOP < 21 mmHg, or, as judged by the physician, target IOP was not reached).

Pseudoexfoliation glaucomas and patients with diabetes were not excluded.

Exclusion Criteria:

All patients in whom beta-blockers were contraindicated were excluded. Ocular Condition.

1. Closed/barely open anterior chamber angles (ACAs) or history of acute angle closure. The ACA was viewed by means of the Goldmann 1-mirror lens. Shaffer grading was used, and grades II, III, and IV were included. Grades 0 and I were excluded.
2. Ocular surgery or argon laser trabeculoplasty within the last 3 months.
3. Ocular inflammation/infection occurring within 3 months before the pretrial visit.
4. Neovascular glaucomas.
5. Hypersensitivity to benzalkonium chloride or to any other component of the trial drug solutions.
6. Other abnormal ocular condition or symptom preventing the patient from entering the trial, according to the investigator's judgement.
7. Patients on either bimatoprost or the LTFC.
8. Patients who had undergone refractive surgery. General
9. Inability to adhere to treatment/visit plan.
10. Participation in any other clinical trial (i.e., requiring in- formed consent) within 1 month before the prestudy visit. 11. Pregnancy, nursing, or, if applicable, nonuse of adequate contraception.

12. Any drug known to affect IOP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Difference in mean diastolic and systolic perfusion pressures | Baseline - Week 2 - Week 6 - Week 12
  The Primary outcome was the difference in mean diastolic and systolic perfusion pressures after bimatoprost and the LTFC

CONTACTS AND LOCATIONS:
Overall Officials: Luca Rossetti, MD, Principal Investigator — A.O. San Paolo Hospital Milan Italy
Locations (9):
- Germany (2):
  - Universitaets-augenklinik, Dresden
  - Universitaets-augenklinik, Magdeburg
- Greece (2):
  - Department of Ophthalmology, University of Thessaly, University Hos- pital of Larissa, Larissa
  - II Department of Ophthalmology, Aristotle University of Thessaloniki, Thessaloniki
- Italy (3):
  - A.O. San Paolo, Milan, Lombardy
  - Clinica Oculistica, Dipartimento di Oftalmologia-Otorinolaringoiatria, Università di Bari, Bari
  - Clinica Oculistica, Università degli studi di Roma, Tor Vergata, Rome
- Universitäts-Augenklinik, Inselspital, University of Bern, Bern, Switzerland
- Moorfields Eye Hospital,, London, United Kingdom

REFERENCES:
- [Result] Rossetti L, Karabatsas CH, Topouzis F, Vetrugno M, Centofanti M, Boehm A, Viswanathan A, Vorwerk C, Goldblum D. Comparison of the effects of bimatoprost and a fixed combination of latanoprost and timolol on circadian intraocular pressure. Ophthalmology. 2007 Dec;114(12):2244-51. doi: 10.1016/j.ophtha.2007.01.025. Epub 2007 Apr 25. PMID 17459480
- [Derived] Rossetti L, Sacchi M, Karabatsas CH, Topouzis F, Vetrugno M, Centofanti M, Boehm A, Vorwerk C, Goldblum D, Fogagnolo P. Comparison of the effects of bimatoprost and a fixed combination of latanoprost and timolol on 24-hour blood and ocular perfusion pressures: the results of a randomized trial. BMC Ophthalmol. 2015 Jan 22;15:7. doi: 10.1186/1471-2415-15-7. PMID 25613811